CLINICAL TRIAL: NCT04177797
Title: A Single Arm Trial of Toripalimab With Neoadjuvant Carboplatin and Paclitaxel for Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Toripalimab With Neoadjuvant Chemotherapy for Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Yongtao Han, Director,Head of Thoracic Surgery, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCH-TS2001
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma; Toripalimab; Neoadjuvant treatment; Chemotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimb (Experimental): Single arm, non randomized, open label study.The patients will receive Toripalimb concurrently caboplatin and paclitaxel treatment.
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Two cycles of Toripalimab(240 mg administered as an intravenous infusion over 30 minutes per 3 weeks), concurrently paclitaxel(135 mg/m2) and carboplatin(AUC 5) administered as an intravenous infusion per 3 weeks.

SUMMARY:
This is a single-institution, single arm trial of Toripalimab with neoadjuvant carboplatin and paclitaxel for locally advanced esophageal squamous cell carcinoma (ESCC).The primary study hypothesis is that the patients who received Toripalimab combined with carboplatin and paclitaxel will increase complete pathologic response rate.

DETAILED DESCRIPTION:
Enrolled patinets will receive two cycles of Toripalimab(240 mg administered as an intravenous infusion over 30 minutes per 3 weeks), paclitaxel(135 mg/m2) and carboplatin(AUC 5) administered as an intravenous infusion per 3 weeks. Giving the drugs on the first day of each cycle.

ELIGIBILITY:
Inclusion Criteria:

* 1.Histologically confirmed ESCC;
* 2.Clinical stage T1-2N2-3M0 or T3N1-3M0 or T4N0-3M0(AJCC 8 TNM classification);
* 3.Have a performance status of 0 or 1 on the ECOG Performance Scale;
* 4.The important organs functions meet the following requirements:the absolute neutrophil count(ANC) ≥1.5×109/L; the platelet count ≥100×109/L; hemoglobin ≥90g/L; bilirubin is less than or equal to 1.5 times ULN, ALT and AST less than or equal 2.5 times UILN; creatinine clearance rate(CCr) ≥50mL/min; the thyroid function is normal;
* 5.Expected survival time is greater than or equal to 3 months;
* 6.Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required;
* 7.Female subjects of childbearing potential must be willing to use an adequate method of contraception - Contraception, for the course of the study through 90 days after the last dose of study medication;
* 8.Be willing and able to provide written informed consent/assent for the trial.

Exclusion Criteria:

* 1.Has any active autoimmune disease or a history of autoimmune disease;
* 2.The patient is receiving systemic steroid therapy or any other form of immunosuppressive therapy;
* 3.The patient had active infection, fever of unknown cause ≥38.5℃ within 7 days before the medication, or white blood cell count at baseline >15×109/L;
* 4.The patient had previously received other anti-pd-1 antibody therapy or other immunotherapy targeting pd-1 / pd-L1,or received chemoradiotherapy;
* 5.Have a history of mental illness or psychiatric substance abuse;
* 6.Patients who had participated in clinical trials of other drugs within 4 weeks;
* 7.Patients with a serious risk to treating patients' safety or a concomitant disease that affects the completion of the study according to the researchers judgment;
* 8.Senior or uncontrolled virus injection: HIV, TP, hepatitis virus;
* 9.Other patients whom the medical practitioner considers inappropriate for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete pathologic response rate | 3 months
  Definition of complete pathologic response is "no cancer cell, including lympho nodes" which corresponds with tumor regression score 0. Definition of pathologic response is as follows. Tumor regression score Grade 0 and 1 will be defined as "responder" and 2 and 3 will be considered as "non-responders"

SECONDARY OUTCOMES:
Disease control rate | 3 months
  According to RECISIST1.1 standard,the disease control rate is the percentage of cases in which relief and stable lesions are obtained after treatment as a percentage of the total evaluable number.
Objective response rate | 3 months
  Objective response rate as assessed by RECISIST1.1 criteria, the percentage of subjects with CR or PR in the total number of subjects in the analysis data set during the period from the beginning of the treatment regimen to the disease progression date.
Incidence of adverse events | 6 months
  Number of participants with treatment-related adverse events as assessed by Number of participants with treatment-related adverse events as assessed by treatment-related adverse events assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China

REFERENCES:
- [Derived] He W, Leng X, Mao T, Luo X, Zhou L, Yan J, Peng L, Fang Q, Liu G, Wei X, Wang K, Wang C, Zhang S, Zhang X, Shen X, Huang D, Yi H, Bei T, She X, Xiao W, Han Y. Toripalimab Plus Paclitaxel and Carboplatin as Neoadjuvant Therapy in Locally Advanced Resectable Esophageal Squamous Cell Carcinoma. Oncologist. 2022 Feb 3;27(1):e18-e28. doi: 10.1093/oncolo/oyab011. PMID 35305102